CLINICAL TRIAL: NCT05139316
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Adeno-Associated Virus Serotype 8-Mediated Gene Transfer of Glucose-6-Phosphatase in Patients With Glycogen Storage Disease Type Ia
Brief Title: A Study of Adeno-Associated Virus Serotype 8-Mediated Gene Transfer of Glucose-6-Phosphatase in Patients With Glycogen Storage Disease Type Ia (GSDIa)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DTX401-CL301; 2020-004184-12 (EudraCT Number); 2023-508750-25-00 (EU CTIS Number)
Record Dates: First submitted 2021-07-14; First posted 2021-12-01 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Glycogen Storage Disease Type IA
Keywords: glycogen storage disorder Ia; AAV; gene therapy; von Gierke disease; glucose metabolism disorder; GSDIa; GSD1
MeSH Terms: conditions — Hepatorenal form of glycogen storage disease; Glycogen Storage Disease Type I; Glucose Metabolism Disorders | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DTX401, Then Placebo (Experimental): Participants receive single peripheral intravenous (IV) infusion of DTX401 in solution. At week 48 participants receive single peripheral IV infusion of Placebo.
  Interventions: Genetic: DTX401; Other: Placebo; Drug: Oral prednisolone; Drug: Placebo for oral prednisolone
- Placebo, Then DTX401 (Placebo Comparator): Participants receive single peripheral IV infusion of Placebo. At week 48 eligible participants receive single peripheral IV infusion of DTX401 solution.
  Interventions: Genetic: DTX401; Other: Placebo; Drug: Oral prednisolone; Drug: Placebo for oral prednisolone
- DTX401 (Japan Only) (Experimental): Participants receive single peripheral intravenous (IV)infusion of DTX401 in solution.
  Interventions: Genetic: DTX401; Drug: Oral prednisolone

INTERVENTIONS:
Genetic: DTX401 — nonreplicating, recombinant, adeno-associated virus (AAV) serotype 8 (AAV8)
  Other Names: pariglasgene brecaparvovec
Other: Placebo — Normal Saline infusion
  Arms: DTX401, Then Placebo; Placebo, Then DTX401
Drug: Oral prednisolone — Participants who receive DTX401 solution will receive oral prednisolone
Drug: Placebo for oral prednisolone — Participants who receive placebo will receive placebo oral prednisolone to maintain the study blind
  Arms: DTX401, Then Placebo; Placebo, Then DTX401

SUMMARY:
The primary objectives of this study are to evaluate the efficacy of DTX401 to reduce or eliminate dependence on exogenous glucose replacement therapy to maintain euglycemia and to maintain or improve the quality of glucose control.

DETAILED DESCRIPTION:
Study DTX401-CL301 is a phase 3 study to determine the efficacy and confirm the safety of DTX401 in patients 8 years and older with glycogen storage disease type Ia (GSDIa).

Participants will be randomized 1:1 to DTX401 or placebo group, and followed closely for 48 weeks. At week 48 eligible participants will cross over and receive DTX401 if they had previously received placebo or placebo if they had previously received DTX401, and will be followed closely for an additional 96 weeks. After completion of week 144 or early withdrawal, participants will be offered enrollment into a Disease Monitoring Program (DMP) where they will be followed for at least 10 years post DTX401 infusion.

In Japan, there will be a single open label study arm and all participants will be treated with DTX401. At week 48, Japanese participants will be offered enrollment into a Disease Monitoring Program (DMP) where they will be followed for at least 10 years post DTX401 infusion.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented GSDIa with confirmation by molecular testing or enzymatic activity on liver biopsy
* Currently receiving a therapeutic regimen of cornstarch (or equivalent), following international guidance/recommendations with stable nutrition, glycemic, and clinical status.
* Willing and able to complete the informed consent process and to comply with study procedures and visit schedule
* Females of childbearing potential and fertile males must consent to use highly effective contraception from the period following informed consent through the duration of the 144-week study and in cases of early withdrawal at least 48 weeks after the last dose of investigational product (IP). Female subjects must agree not to become pregnant. Male subjects must agree not to father a child or donate sperm

Key Exclusion Criteria:

* Detectable pre-existing antibodies to the AAV8 capsid
* History of liver transplant, including hepatocyte cell therapy/ transplant
* History of liver disease
* Presence of liver adenoma >5 cm in size
* Presence of liver adenoma >3 cm and ≤5 cm in size that has a documented annual growth rate of ≥0.5 cm per year
* Significant hepatic inflammation or cirrhosis as evidenced by imaging or any of the following laboratory abnormalities: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > upper limit of normal (ULN), total bilirubin >1.5 × ULN, alkaline phosphatase >2.5 × ULN
* Non-fasting triglycerides ≥1000 mg/dL
* Pregnant, breastfeeding, or planning to become pregnant (self or partner) at any time during the study.
* Current or previous participation in another gene transfer study
* History of illicit drug use within 60 days prior to screening or positive results from an 8-panel urine drug screen during the Screening Period completed at 2 time points at least 4 weeks apart

Note: additional inclusion/exclusion criteria may apply, per protocol

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline to Week 48 in Daily Cornstarch Intake | Baseline, Week 48

SECONDARY OUTCOMES:
Change from Baseline to Week 48 in Number of Total Daily Doses of Cornstarch in DTX401 Group Compared to Placebo Group | Baseline, Week 48
Change from Baseline to Week 48 in Percentage of Glucose Values in Hypoglycemic Range (<70mg/dL [3.9 mmol/L]) | Baseline, Week 48
Patient Global Impression of Change (PGIC) Assessment Score at Week 48 | Baseline, Week 48
Change from Baseline to Week 48 in Time to Hypoglycemia (<54 mg/dL [3.0 mmol/L]) During a Controlled Fasting Challenge | Baseline, Week 48
Change from Baseline to Week 48 in Percentage of Glucose Values in the Range of 70-120 mg/dL (3.9-6.7 mmol/L) | Baseline, Week 48
Number of Treatment Emergent Adverse Events (TEAEs), TEAEs of Special Interest, Serious TEAEs, Related TEAEs, Discontinuations From Study or Investigational Product Due to Adverse Events (AEs), and Fatal AEs | up to 144 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (20):
- United States (9):
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Mount Sinai, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil
- McGill University, Montreal, Quebec, Canada
- Righospitalet, Copenhagen, Capital, Denmark
- University Medical Center Eppendorf, Hamburg, Germany
- Italy (2):
  - Istituto Giannina Gaslini, Genova, Linguria
  - University of Naples, Naples
- Japan (3):
  - Kumamoto University Hospital, Kumamoto
  - Osaka City General Hospital, Osaka
  - Fujita Health University Hospital, Toyoake
- Groningen University, Groningen, Netherlands
- Hospital Clinico Universitario de Santiago, Santiago de Compostela, A Coruna, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultragenyx Patient Advocacy/GSDIA Disease Information — https://ultrarareadvocacy.com/conditions-we-study/glycogen-storage-disease-type-ia-gsdia/
- See also: Ultragenyx Transparency Commitment — http://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/